CLINICAL TRIAL: NCT00232765
Title: A Multicenter, Randomized, Double-Blind Study of the Sirolimus-Coated BX VELOCITYTM Balloon-Expandable Stent in the Treatment of Patients With de Novo Coronary Artery Lesions
Brief Title: Study of Sirolimus-Coated BX VELOCITY Balloon-Expandable Stent in Treatment of de Novo Native Coronary Artery Lesions (SIRIUS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sid Cohen, MD, PhD, Cordis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P00-6302
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cypher Bx Velocity
  Interventions: Device: CYPHER Sirolimus-Eluting Stent
- 2 (Active Comparator): Uncoated Bx Velocity
  Interventions: Device: Uncoated BX VELOCITY Balloon-Expandable Stent

INTERVENTIONS:
Device: CYPHER Sirolimus-Eluting Stent — CYPHER Sirolimus-Eluting Stent
  Arms: 1
Device: Uncoated BX VELOCITY Balloon-Expandable Stent — Uncoated BX VELOCITY Balloon-Expandable Stent
  Arms: 2

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the sirolimus-coated Bx VELOCITYTM stent in reducing target vessel failure in de novo native coronary artery lesions as compared to the uncoated Bx VELOCITYTM balloon-expandable stent. Both stents are mounted on the Raptorâ over-the-wire (OTW) Stent Delivery System.

DETAILED DESCRIPTION:
This is a multicenter (55 sites), prospective, 2-arm randomized, double-blind study designed to assess the safety and effectiveness of the sirolimus-coated Bx VELOCITYTM stent as compared to the uncoated Bx VELOCITYTM stent. A total of 1100 patients will be entered in the study and will be randomized on a 1:1 basis. Patients with de novo native coronary artery lesions >/=15mm and </=30mm in length and >/=2.50mm to </=3.5mm in diameter by visual estimate who meet all eligibility criteria will be either randomized to the sirolimus-coated Bx VELOCITYTM stent or the uncoated Bx VELOCITYTM stent. Patients will be followed at 30 days, 3, 6, 9 and 12 months, and 2, 3, 4, 5, 6, 7, and 8 years post-procedure, with approximately 850 patients having repeat angiography at 8 months. A subset of approximately 17 centers will participate in an intravascular ultrasound (IVUS) sub study, in which all patients at these centers will be enrolled in the sub study. Additionally, data will be collected for a medical economic analysis. These data will include costs associated with the index hospitalization and length of stay, and rehospitalizations during the 12-month follow-up period. This is a single lesion treatment study. Patients who have had interventions of other lesions within 30 days of the study procedure or have interventions planned after the index procedure are excluded. It is anticipated that the total length of the study will be 101 months: 5 months to complete patient enrollment and 8 years for follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female patients minimum 18 years of age
2. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II) OR patients with documented silent ischemia;
3. Target lesion is 2.50mm and 3.5mm in diameter (visual estimate);
4. Target lesion is 15mm and 30mm in length (visual estimate);
5. Target lesion stenosis is >50% and <100% (visual estimate);

Exclusion Criteria:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK >2 times normal within the preceding 24 hours and the CK and CK-MB enzymes remains above normal at the time of treatment;
2. Has unstable angina classified as Braunwald III B or C, or is having a peri infarction;
3. Documented Left ventricular ejection fraction 25%;
4. Impaired renal function (creatinine > 3.0 mg/dl) at the time of treatment;
5. Target lesion involves bifurcation including a diseased side branch 2.5mm in diameter (either stenosis of both main vessel and major branch or stenosis of just major branch) that would require treatment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1058 (Actual)
Dates: Start 2001-02; Primary Completion 2002-05 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Target vessel failure (TVF) defined as cardiac death, myocardial infarction, or target vessel revascularization at 9 months post-procedure. | 9 months post procedure

SECONDARY OUTCOMES:
Composite of MACE defined as death, myocardial infarction (Q wave and non-Q wave), emergent bypass surgery, or repeat target vessel revascularization at 30 dys and 3, 6, 9, and 12 mo, and 2, 3, 4, 5, 6, 7, and 8 yrs post-procedure; | 30 dys and 3, 6, 9, and 12 mo, and 2, 3, 4, 5, 6, 7, and 8 yrs post-procedure
Angiographic binary restenosis (>/=50% diameter stenosis) 8 mo post-procedure; | 8 months post-procedure
In-stent and in-lesion MLD at 8 mo post-procedure; | 8 months post-procedure
Target lesion revascularization at 9 mo post-procedure; | 9 months post-procedure
Target vessel revascularization at 9 mo post-procedure; | 9 months post-procedure
Device success defined as achievement of a final residual diameter stenosis of <50% (by QCA), using the assigned device only. If QCA is not available, the visual estimate of diameter stenosis is used; | Study Completion
Lesion success defined as the attainment of <50% residual stenosis (by QCA) using any percutaneous method; | Study Completion
Procedure success defined as achievement of a final diameter stenosis of <50% (by QCA) using any percutaneous method, without the occurrence of death, MI, or repeat revascularization of the target lesion during the hospital stay; | During the hospital stay
Costs associated with the index hospitalization and length of stay, and repeat hospitalizations during the 12-month post-procedure follow-up period. | 12-month post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Martin B. Leon, MD, Principal Investigator — New York Presbyterian Hospital/Columbia University Medical Center; Jeffrey Moses, MD, Principal Investigator — New York Presbyterian Hospital/Columbia University Medical Center
Locations (1):
- New York Presbyterian Hospital/Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Result] Weisz G, Leon MB, Holmes DR Jr, Kereiakes DJ, Popma JJ, Teirstein PS, Cohen SA, Wang H, Cutlip DE, Moses JW. Five-year follow-up after sirolimus-eluting stent implantation results of the SIRIUS (Sirolimus-Eluting Stent in De-Novo Native Coronary Lesions) Trial. J Am Coll Cardiol. 2009 Apr 28;53(17):1488-97. doi: 10.1016/j.jacc.2009.01.050. PMID 19389558
- [Result] Popma JJ, Tiroch K, Almonacid A, Cohen S, Kandzari DE, Leon MB. A qualitative and quantitative angiographic analysis of stent fracture late following sirolimus-eluting stent implantation. Am J Cardiol. 2009 Apr 1;103(7):923-9. doi: 10.1016/j.amjcard.2008.12.022. PMID 19327417
- [Result] Chacko R, Mulhearn M, Novack V, Novack L, Mauri L, Cohen SA, Moses J, Leon MB, Cutlip DE. Impact of target lesion and nontarget lesion cardiac events on 5-year clinical outcomes after sirolimus-eluting or bare-metal stenting. JACC Cardiovasc Interv. 2009 Jun;2(6):498-503. doi: 10.1016/j.jcin.2009.03.013. PMID 19539252
- [Derived] Spaulding C, Daemen J, Boersma E, Cutlip DE, Serruys PW. A pooled analysis of data comparing sirolimus-eluting stents with bare-metal stents. N Engl J Med. 2007 Mar 8;356(10):989-97. doi: 10.1056/NEJMoa066633. Epub 2007 Feb 12. PMID 17296825